CLINICAL TRIAL: NCT05869227
Title: The Efficacy and Safety of Maintenance Therapy With Toripalimab Combined With Capecitabine/Placebo for Recurrent and Metastatic Nasopharyngeal Carcinoma:Randomized, Double-blind, Placebo-controlled, Multicenter Phase III Clinical Study
Brief Title: Maintenance Therapy With Toripalimab Combined With Capecitabine/Placebo for Recurrent and Metastatic Nasopharyngeal Carcinoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: XIANG YANQUN (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Zhujiang Hospital (Other)
Responsible Party: Sponsor-Investigator, XIANG YANQUN, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SYSKY-2023-307-02
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Nasopharyngeal Carcinoma; Maintenance Therapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Capecitabine; toripalimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capecitabine combined with toripalimab maintenance group (Experimental): Capecitabine, 1000 mg/m2/dose, twice a day, days 1-14; 21 days/cycle toripalimab, 240mg, intravenously, day 1 and 21 days/cycle
  Interventions: Drug: Capecitabine/Placebo combined with toripalimab
- Placebo combined with toripalimab maintenance group (Placebo Comparator): Placebo, 1000 mg/m2/dose, twice a day, days 1-14; 21 days/cycle toripalimab, 240mg, intravenously, day 1 and 21 days/cycle
  Interventions: Drug: Capecitabine/Placebo combined with toripalimab

INTERVENTIONS:
Drug: Capecitabine/Placebo combined with toripalimab — Combined

SUMMARY:
The aim of this study is to investigate the efficacy and safety of the "capecitabine combined with toripalimab maintenance regimen" in improving the first-line treatment of recurrent and metastatic nasopharyngeal carcinoma after receiving remission through chemotherapy combined with anti PD-1 monoclonal antibody standard regimen.

ELIGIBILITY:
Inclusion Criteria:

1. The age at the time of diagnosis is 18-75 years old, regardless of gender;
2. Histologically confirmed nasopharyngeal carcinoma;
3. Confirm the presence of distant metastasis in advanced nasopharyngeal carcinoma patients or recurrent nasopharyngeal carcinoma patients who cannot receive local treatment. ;
4. After receiving standard treatment for 4-6 cycles, the disease is control;
5. ECOG score 0-1;
6. Expected survival time of at least 12 weeks;
7. Patients who have not received systemic chemotherapy within 6 months prior to diagnosis ;
8. According to RECIST 1.1 standard, at least 1 measurable lesion;
9. Enough organ function;
10. Sign an informed consent form;
11. Female participants with fertility and male participants with fertility partners must agree to use reliable contraceptive measures within 6 months after screening and the last treatment.

Exclusion Criteria:

1. Patients who are known to be intolerant to capecitabine or allergic to any therapeutic drug, or who are participating in clinical studies of other new drugs;
2. Diseases that may interfere with oral medication treatment, including but not limited to swallowing difficulties, chronic diarrhea, or intestinal obstruction;
3. Previous or current history of other tumors, excluding cured cervical carcinoma in situ, skin basal cell carcinoma, and thyroid papillary carcinoma;
4. Sever heart disease;
5. Central nervous system metastasis with clinical symptoms;
6. Serious infections ;
7. Within 4 weeks of signing the informed consent form, receive systemic hormone or other immunosuppressive therapy with an equivalent dose greater than 10mg prednisone per day. Subjects with a systemic hormone dose ≤ 10mg prednisone per day or inhaled/topical corticosteroids can be enrolled in the study;
8. Patients with active chronic hepatitis B or active hepatitis C.
9. A history of interstitial pneumonia or other autoimmune diseases.
10. HIV infection;
11. Individuals with significant organ dysfunction or uncontrollable comorbidities, including but not limited to uncontrollable hypertension, decompensated liver cirrhosis, active peptic ulcer, or hemorrhagic disease;
12. Less than 6 weeks after major organ surgery;
13. Pregnant or breast feeding;
14. Patients with mental illness, those with a history of alcohol or drug abuse, or those who are unable to obtain informed consent;
15. Other researchers have determined that it is not suitable to participate in this trial.
16. Those who refuse or are unable to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2027-12-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2 years
  Progression free survival is defined as the time interval between randomization and the first recording of tumor progression (evaluated according to RECIST 1.1 criteria, regardless of continued treatment) or death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- SunYat-senU, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No